CLINICAL TRIAL: NCT03254706
Title: Effect of Increased Improve Time on Adhesive System: A RANDOMIZED CLINICAL TRIAL
Brief Title: Effect of Increased Improve Time on Adhesive System
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Ponta Grossa (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Eloisa Andrade de Paula, Doctor, Universidade Estadual do Oeste do Paraná
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 57317816.6.0000.5084
Record Dates: First submitted 2017-08-15; First posted 2017-08-18 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Clinical Trial
Keywords: Dentin adhesive; Non-carious cervical lesions; Longevity.
MeSH Terms: interventions — 1,2-dihydroxy-4-(nitroethenyl)benzene

STUDY DESIGN:
Intervention Model Description: This was a double-blind, superiority, split-mouth randomized clinical trial. The study was carried out in the clinics of the School of Dentistry at the local University from August 2015 to August 2017.
Who Masked: Participant, Outcomes Assessor
Masking Description: A staff member not involved in the research protocol performed the randomization process with computer-generated tables. Details of the allocated groups were recorded on cards contained in sequentially numbered, opaque, sealed envelopes. Opening the envelope only on the day of the restorative procedure guaranteed the concealment of the random sequence. The examiners were not involved with the restoration procedures and therefore blinded to the group assignment, performed the clinical evaluation. Patient were also blinded to group assignment in a double-blind randomized clinical trial design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Peak etch-and-rinse (P1) (Active Comparator): Application Mode - According to the manufacturer's instructions.
  Interventions: Other: Peak etch-and-rinse (P1)
- Peak applied for double time(P2X) (Experimental): Application Mode - According to the manufacturer's instructions, but for the double time.
  Interventions: Other: Peak applied for double time(P2X)
- Single Link etch-and-rinse (SL1) (Active Comparator): Application Mode - According to the manufacturer's instructions.
  Interventions: Other: Single Link etch-and-rinse (SL1)
- Single Link double time (SL2X) (Experimental): Application Mode - According to the manufacturer's instructions, but for the double time.
  Interventions: Other: Single Link double time (SL2X)

INTERVENTIONS:
Other: Peak etch-and-rinse (P1) — Application Mode - Peak Adhesive system applied according to the manufacturer's instructions.
  Other Names: P1
  Arms: Peak etch-and-rinse (P1)
Other: Peak applied for double time(P2X) — Application Mode - Peak Adhesive system applied according to the manufacturer's instructions, but for the double time.
  Other Names: P2X
  Arms: Peak applied for double time(P2X)
Other: Single Link etch-and-rinse (SL1) — Application Mode - Single Link Adhesive system applied according to the manufacturer's instructions.
  Other Names: SL1
  Arms: Single Link etch-and-rinse (SL1)
Other: Single Link double time (SL2X) — Application Mode - Single Link Adhesive system applied according to the manufacturer's instructions, but for the double time.
  Other Names: SL2X
  Arms: Single Link double time (SL2X)

SUMMARY:
Objective: This double-blind randomized clinical trial evaluates the influence of increased application time of a new etch-and-rinse two-step adhesive Single Link; (Angelus Dental Products Industry) applied in non-carious cervical lesions (NCCLs).

Methods: A total of 221 restorations were randomly placed in 35 patients assigned in four groups to two different etch-and-rinse two-step adhesive Peak® Universal Bond (P) (Ultradent Products Ind) and Single Link (SL) (Angelus Dental Products Industry). The adhesives systems were applied on the NCCLs follows: P1 - applied according to the manufacturer's; P2X - applied for the double time; SL1 and; SL2X. The resin composite Amelogen (Ultradent) was placed incrementally. The restorations were evaluated imediataly (baseline), 6 and 12 months, using the FDI and USPHS criteria. Statistical analyses were performed using appropriate tests (=0.05).

DETAILED DESCRIPTION:
Methods:

Recruitment Patients were recruited as they seek for treatment in the clinics of Dentistry of the local university. No advertisement was made for participant recruitment. Patients were recruited in the order in which they reported for the screening session, thus forming a sample of convenience.

Eligibility criteria A total of 183 participants were examined by two calibrated dental students to check if they met the inclusion and exclusion criteria.

Sample size calculation The annual retention rate to one-step self-etch adhesives in NCCLs was reported to be 4.4% in a recent systematic review. Considering that this decline follow a linear trend, the overall retention rate of one-step self-etch adhesives will be approximately 78% after 5-year of clinical service. With an of 0.05, a power of 80%, and a two-sided test, the minimal sample size will be 41 restorations in each group in order to detect a difference of equivalence of 15% among the test groups.

Interventions A total of 221 restorations were randomly placed in 35 patients assigned in four groups to two different etch-and-rinse two-step adhesive Peak® Universal Bond (P) (Ultradent Products Ind) and Single Link (SL) (Angelus Dental Products Industry).

The adhesives systems were applied on the NCCLs follows: P1 - applied according to the manufacturer's; P2X - applied for the double time; SL1 and; SL2X. The resin composite Amelogen (Ultradent) was placed incrementally. The restorations were evaluated imediataly (baseline), 6 and 12 months, using the FDI and USPHS criteria. Statistical analyses were performed using appropriate tests (=0.05).

ELIGIBILITY:
Inclusion Criteria:

Participants had to be in good general health, at least 18 years old, have an acceptable oral hygiene level, and present at least 20 teeth under occlusion, at least four NCCLs in four different teeth, these lesions had to be non-carious, non-retentive, deeper than 1 mm, and involve both the enamel and dentin of vital teeth without mobility. The cavo-surface margin could not involve more than 50% of enamel, and all lesions had cervical margins ending in dentin.

Exclusion Criteria:

Participants had not be in good general health, at less 18 years old, have not an acceptable oral hygiene level, and present at less 20 teeth under occlusion, at less four NCCLs in four different teeth, these lesions had not be non-carious, retentive and involve only enamel of vital teeth with mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Retention/fracture | 6 months
  The primary clinical endpoint was restoration retention/fracture

SECONDARY OUTCOMES:
Marginal staining | 6 months
  restoration Marginal staining
marginal adaptation | 6 months
  restoration marginal adaptation
postoperative sensitivity | 6 months
  restoration postoperative sensitivity
recurrence of caries. | 6 months
  restauration recurrence of caries

CONTACTS AND LOCATIONS:
Overall Officials: Márcio Camargo, Master, Study Chair — Universidade Estadual do Oeste do Paraná
Locations (1):
- Universidade Estadual do Oeste do Paraná, Cascavel, Paraná, Brazil